CLINICAL TRIAL: NCT04165941
Title: A Phase I Study of Drug Resistant Immunotherapy (DRI) With Activated, Gene Modified γδ T Cells in Patients With Newly Diagnosed Glioblastoma Multiforme Receiving Maintenance Temozolomide Chemotherapy
Brief Title: Novel Gamma-Delta (γδ)T Cell Therapy for Treatment of Patients With Newly Diagnosed Glioblastoma
Acronym: DRI
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Louis Burt Nabors, MD, Professor, Neurology Chair Office, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UAB 1773
Record Dates: First submitted 2019-11-12; First posted 2019-11-18 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Brain Tumor Adult
Keywords: Newly diagnosed brain tumor; Phase 1; Drug Resistant Immunotherapy; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- DRI cell therapy (Experimental): The only arm will receive the DRI modified gamma delta T cells following standard therapy with radiation and temozolomide chemotherapy concurrent.
  Interventions: Biological: DRI cell therapy

INTERVENTIONS:
Biological: DRI cell therapy — Drug Resistant Immunotherapy with gamma delta modified T cells to be resistance to temozolomide will be infused into the surgical cavity following the completion of standard concurrent radiation and chemotherapy with temozolomide.

SUMMARY:
This study is being conducted to find out if the safety and tolerability of an experimental cell therapy is safe to administer to patients with a newly diagnosed glioblastoma multiforme (GBM) in combination with temozolomide (TMZ).

DETAILED DESCRIPTION:
The cell therapy that is being used in this study is called gene-modified gamma delta T cells or Drug Resistant Immunotherapy (DRI). Gamma delta T cells are a type of lymphocyte or white blood cell that may help the immune system to recognize and kill cancer cells. Some chemotherapy can kill these gamma delta T cells. For the cell therapy being used in this study, the genes or DNA within these gamma delta T cells are modified so they are resistant to or may not be affected by chemotherapy. The chemotherapy that is being used in this study is called temozolomide (TMZ) and can reduce the number of these gamma delta T cells or lymphocytes. This study will also find out if these modified gamma delta T cells (DRI) are unaffected by TMZ. The DRI is given in combination with a standard dose of TMZ and is administered into the brain where the tumor is located.

After subjects are consented in Parts A and B of the study, approximately about 2 tablespoons of blood will be collected for tests that may provide additional information about subjects T cells and how they may respond to treatment.

Part A Subjects will have a surgical procedure completed that will remove their tumor (called a surgical resection). They will have a Rickham catheter placed which is a device typically used to deliver chemotherapy into the brain. The infusion catheter will be placed first prior to the tumor resection. A sample of tumor tissue will be taken and examined to confirm the diagnosis of GBM. The diagnosis of GBM must be confirmed prior to beginning Part B.

Part B After the surgical resection and on Study Day 1, subjects will return to the study doctor's office/clinic to undergo a procedure called apheresis. This procedure will separate out cells called peripheral blood mononuclear cells (PBMC). Apheresis is the removal of blood plasma from the body by collecting your blood and separating the plasma from the PBMCs. These cells include the gamma delta T cells that will be used to synthesize the DRI γδ T cells. Once the cells for the DRI γδ T cells are synthesized, they are reintroduced into subject's brain through the Rickham catheter.

Following apheresis and confirmation that the required number of gamma delta T cells were collected, subjects will begin the recommended or standard of care treatment for newly diagnosed GBM. This will include 6 weeks of chemotherapy with TMZ and radiation. Subjects will then have about 4 weeks of no treatment prior to beginning the Part B maintenance phase of treatment, which includes 6 cycles of TMZ. Depending on which dose level they receive, they will be administered either 1 injection of the DRI γδ T cells or 3 and these will be injected through the Rickham catheter.

The first 3 subjects will receive a single dose of the DRI γδ T cells at the lowest dose level. Subjects receiving a single dose of the DRI γδ T cells will be observed for a of minimum 30 days from the time the first subject is enrolled, followed by a minimum of 7 days between each additional subject enrolled to allow for evaluation of potential side effects. If the DRI γδ T cell injection does not cause serious side effects, the second set of 3 subjects will be enrolled. The second set of 3 patients will receive 3 doses of the DRI γδ T cells. The approximate duration of the study may be up to 15 years, or until disease progression or subjects withdraw from the study.

ELIGIBILITY:
Inclusion Criteria:

* Must have magnetic resonance imaging (MRI) features consistent with and suspicious for malignant glioma. This will be Part A - Tissue (biopsy) and Rickham catheter placement.
* Must have histologically or cytologically confirmed glioblastoma multiforme prior to administration of the DRI γδ T cell injection. This will be Part B - Screening and Study Treatment.
* Prior therapy: Must have completed a standard temozolomide and radiotherapy treatment as described in Part A and be eligible to receive maintenance therapy with temozolomide (consistent with NCCN guidelines for newly diagnosed GBM and maintenance therapy).
* Age ≥18 yearsΦ: Because no dosing or adverse event data are currently available on the use of γδ T cells in patients <18 years of age, children are excluded from this study but will be eligible for future pediatric Phase I single-agent trials.
* Karnofsky Performance Status ≥70%
* Life expectancy of greater than 12 weeks
* Patients must have organ and marrow function as defined below:

  1. leukocytes >3,000/µl
  2. absolute neutrophil count >1,500/µl
  3. Hgb greater than or equal to 9.0 g/dL
  4. platelets >100,000/µl
  5. total bilirubin within normal institutional limits
  6. AST (SGOT)/ALT (SGPT) <2.5 X institutional upper limit of normal
  7. Normal electrolyte levels including sodium, calcium, potassium, chloride and magnesium
  8. INR/PT/aPTT ≤1.5xULN
  9. Normal EKG; if abnormal, NCS
  10. Normal blood presure as adjusted for age
* Creatinine within normal institutional limits or if higher than the normal range, calculated creatinine clearance (CrCl) must be ≥ 50 mL/min/1.73 m2 (e.g., by Cockcroft-Gault formula); actual body weight must be used for CrCl unless body mass index (BMI) is > 30 kg/m2, in which case, lean body weight must be used

Exclusion Criteria:

* Patients who have received any therapy for the treatment of GBM prior to inclusion in Part A and any treatment other than standard of care as described in Part A of this study including: cellular immunotherapy or gene therapy within 6 weeks prior to entering the study, surgical resection or alkylating agent chemotherapy within 4 weeks prior to entering the study, or have received experimental immunotherapy at any time, and those who have not recovered from adverse events due to therapeutic interventions administered more than 4 weeks earlier.
* Patients may not be receiving any other investigational agents.
* Contraindication to the placement of an intracranial access device (Rickham catheter) at the time of surgery.
* Prior history of encephalitis, multiple sclerosis, or other CNS infection
* Required steroid increase within 2 weeks of scheduled DRI γδ T cells administration.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or any othermedical condition that precludes surgery. Also, psychiatric illness/social situations that would limit compliance with study requirements.
* Allergies/hypersensitivity: Aminobisphosphonates such as Zoledronate®, Pamidronate® or similar
* Pregnant women are excluded from this study because the lentiviral- modified γδ T cells designed to express MGMT cells have an unknown potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with these cells, breastfeeding should be discontinued if the mother is treated with the lentiviral-modified γδ T cells designed to express MGMT. The following birth control methods are acceptable for this study in women of child- bearing potential:
* A Combination of TWO of the following:

  1. Barrier method of contraception:

     1. condoms (male or female) with or without a spermicidal agent, diaphragm or cervical cap with spermicide
     2. IUD
  2. Hormone-based Contraceptive
* Note: Drug-drug interactions with some ARVs will make hormonal contraception a less reliable method.
* Because patients with immune deficiency will be unable to mount the anticipated immune response underlying this therapeutic rationale, HIV-seropositive patients are excluded from this study.
* Some of the contraceptive methods listed above may not prevent the spread of HIV to other people. Patients should discuss their contraceptive choices with their health care provider to choose the best way to both prevent pregnancy as required by this study and to prevent the spread of HIV to any partner(s).
* Patients with history of prior organ or bone marrow transplantation are not eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-02-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary: Highest safe dose frequency or maximally planned dose, if no dose-limiting toxicity observed. | 12 weeks
  Safety and toxicity of intracranially infused DRI gamma delta T cells

SECONDARY OUTCOMES:
Time to progression | Through study completion, on average one year
  Time to disease progression
Overall survival | Through study completion, on average one year
  Time that participants survive
Assessment of biological activity | Through study completion, on average one year
  Serum measurements of cell therapy activity

CONTACTS AND LOCATIONS:
Overall Officials: Louis B Nabors, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nabors LB, Lamb LS, Goswami T, Rochlin K, Youngblood SL. Adoptive cell therapy for high grade gliomas using simultaneous temozolomide and intracranial mgmt-modified gammadelta t cells following standard post-resection chemotherapy and radiotherapy: current strategy and future directions. Front Immunol. 2024 Feb 7;15:1299044. doi: 10.3389/fimmu.2024.1299044. eCollection 2024. PMID 38384458
- [Derived] Zhao Y, Dong P, He W, Zhang J, Chen H. gammadelta T cells: Major advances in basic and clinical research in tumor immunotherapy. Chin Med J (Engl). 2024 Jan 5;137(1):21-33. doi: 10.1097/CM9.0000000000002781. Epub 2023 Aug 18. PMID 37592858